CLINICAL TRIAL: NCT03642678
Title: Intervention Study for Validation of Application of a Prediction Model in Maintenance Hemodialysis Patients
Brief Title: Dialysis Model for Outcome and Nutrition Decision
Acronym: DIAMOND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: An Hsin QingShui Clinic (Other)
Responsible Party: Principal Investigator, Chen Huan Sheng, Principal Investigator, An Hsin QingShui Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DIAMOND
Record Dates: First submitted 2018-08-18; First posted 2018-08-22 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Protein-Calorie Malnutrition
Keywords: Prediction Model; Malnutrition; Hemodialysis
MeSH Terms: conditions — Protein-Energy Malnutrition; Malnutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants identified as high-risk for malnutrition-related mortality by prediction model are cluster-randomized into study group.
  Interventions: In this group, participants will be given common clinical screening for clinical or sub-clinical infection and also oral nutrition supplement (ONS) if albumin is < 3.8 g/dl. Parameters for outcome measurements are recorded monthly (such as biochemical data) or quarterly (such as Body Composition Monitor (BCM) or Malnutrition Inflammatory Score (MIS). Hospitalization or Mortality events will be recorded when happened.
  Interventions: Dietary Supplement: ONS
- Control group (No Intervention): Participants identified as high-risk for malnutrition-related mortality by prediction model are cluster-randomized into control group. In this group, participants will not be given any intervention, but only outcome measurements are recorded monthly (such as biochemical data) or quarterly (such as Body Composition Monitor (BCM) or Malnutrition Inflammatory Score (MIS). Hospitalization or Mortality events will be recorded when happened.

INTERVENTIONS:
Dietary Supplement: ONS — High-risk patients identified by prediction model in study group are intervened by pre-defined intervention protocol, which include oral nutrition supply, infection prevention, bp control and improving of dialysis therapy options and so on.
  Other Names: Clinical Infection Screening; Clinical procedure for malnutrition prevention
  Arms: Intervention group

SUMMARY:
This study is the secondary phase of Taiwan Prediction Model Project Plan (TPMPP). The investigators try to design a prospective randomized control trial with nutrition intervention to validate 3 prediction models the investigators developed in the first phase. Proper validation of these models is mandatory before they can be applied and implemented into daily clinical practice. At present, around 20 centers with estimated around 550-650 high-risk patients will be enrolled with 1:1 ratio in study and control groups. Following up of parameters about primary and secondary outcomes will be done in both groups. But a pre-designed intervention protocol, which is according to 3 elucidated screening methods, will be applied only to the study group. The total study period will be one year.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a major public health concern. Progression of CKD leads to end-stage renal disease (ESRD), a total and permanent failure of kidney function requiring kidney transplant or maintenance hemodialysis. Among the numerous risk factors of mortality, severe malnutrition, now defined as protein energy wasting (PEW), which is manifested by low serum levels of albumin or pre-albumin, sarcopenia and weight loss, is one of the strongest predictors of mortality, morbidity and infection-related hospitalizations in hemodialysis (HD) patients. When PEW is present or the patient is at high risk, oral intradialytic or daily supplements, aiming at increasing energy and protein intake, while in selected cases intra-dialytic parenteral nutrition may be used for the clinician. Previous reports showed that providing patients with intradialytic food, liquid supplements, or parenteral nutrition has been shown to compensate for this loss. In patients with ESRD, it is important to prevent PEW through a regular nutritional status evaluation and nutritional counseling by a renal dietitian. Intradialytic administration of oral or parenteral supplementation of nutrients is safe and should be encouraged in selected patients. Although the problem of malnutrition became more and more serious due to the increasingly aging and Diabetes Mellitus (DM) proportion in HD population, there are still no universally accepted methods to early detect or predict this problem. Thus, the intention for early intervention to suitable patients faces difficulty. In Taiwan Prediction Model Project Plan (TPMPP), the investigators try to develop a model using common available clinical data with the utilization of current machine learning methods to early detect the patients with high risks for malnutrition and the investigators wish through the routine application of this model, the investigators can do nutrition intervention in much earlier stage and improve the patients' outcome. In the first stage of TPMPP, the investigators have developed some prediction models through an abundant retrospective database collected in Fresenius Database (NephroWeb) from 2011-2018. Before real implementation of these models in clinical practice, the investigators need to validate these models with prospective design with proper intervention, this is the main purpose of this study. The Body Composition Monitor with the principle of Bioimpedance Spectroscopy (BCMBIS, Fresenius Medical Care) is a simple and accurate tool for the assessment of body composition. Recently, the lean and fat mass indexes (LTI, FTI), derived from BCM, have become good predictors of mortality in HD individuals, which have been more sensitive to malnutrition, and altogether anthropometric indicators may result in an early detection of mortality risk in this population. Thus, the investigators also try to apply these parameters in this study as important nutrition outcomes for follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Maintenance Hemodialysis Patients (MHD) patients from multiple centers identified by the risk models as high-risk patients

Exclusion Criteria:

* Acute patients
* Terminal Cancer Patients with life expectancy < 3 months
* Age < 20 year-old
* Active infection, including Tuberculosis and AIDS
* Patients received ONS 1 month before enrollment
* Pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 422 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2022-04-26 (Actual)

PRIMARY OUTCOMES:
1-year mortality | up to 12 months
  1-year mortality evaluated by cox model and logistic regression

SECONDARY OUTCOMES:
Serum Albumin concentration change | up to 12 months
  comparing the serum albumin concentration in intervention and control groups during study.

CONTACTS AND LOCATIONS:
Overall Officials: Huan Sheng Chen, MD, Principal Investigator — An Hsin QingShui Clinic
Locations (1):
- An Hsin Clinic, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No